CLINICAL TRIAL: NCT01173679
Title: Phase II Trial of Dasatinib With Fludarabine and Rituximab in Relapsed and Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Brief Title: Dasatinib With Fludarabine and Rituximab in Relapsed and Refractory CLL and SLL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Philip C. Amrein, M.D., Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-325
Record Dates: First submitted 2010-07-28; First posted 2010-08-02 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CLL; fludarabine; rituximab; dasatinib; refractory; relapsed
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Dasatinib; Rituximab; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dasatinib, rituximab, fludarabine (Other): Single-arm, open-label
  Interventions: Drug: dasatinib; Drug: Rituximab; Drug: fludarabine

INTERVENTIONS:
Drug: dasatinib — Taken orally once a day on days 1-14 of each 28-day cycle
Drug: Rituximab — Given intravenously, 375 mg/m2 each cycle (dose split, given on Days 3+4 of cycle 1, variable after that).
Drug: fludarabine — Given intravenously, 25 mg/m2/day, for 3 doses per cycle (Days 3-5 in cycle 1, Days 1-3 after that)

SUMMARY:
Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL) are similar diseases of the white blood cells and are typically treated the same way. Recent research shows that a key enzyme in CLL cells is responsible for cell survival. This enzyme is called LYN kinase. Laboratory studies show that inhibition of LYN kinase in CLL cells results in the death of CLL cells. Dasatinib has the ability to inhibit LYN kinase and, therefore, should have some effect on CLL cells. The purpose of this study is to see of the study drug dasatinib, in combination with fludarabine and rituximab, is safe and effective to use for people with relapsed or refractory CLL/SLL.

DETAILED DESCRIPTION:
* Since the purpose of the study is to determine the response rate of the 3 drug regimen, everyone who participates will receive the same dose of the study drug, dasatinib and the 2 standard drugs, fludarabine and rituximab.
* Participants will receive the drugs dasatinib, fludarabine, and rituximab at the following time points through each cycle of treatment. A cycle of study treatment is 28 days. Dasatinib pills will be taken orally each day for the first 2 weeks of each cycle. Fludarabine will be give intravenously on three days of each cycle (Days 3-5 in the first cycle, days 1-3 after that). Rituximab will be given intravenously with a total dose of 375 mg/m2 each cycle (split on Days 3+4 in the first cycle and at the discretion of the treating physician after that on Days 1-3).
* The following procedures will be repeated throughout the study: medical history review; physical exam; performance status test; blood tests and EKG. They will occur daily during the first week of treatment, then weekly for the rest of cycle 1. After cycle 1 these procedures will be done once a week for 4 weeks then once a month for 6 months.
* Tumor assessments will be repeated once every 2 months for the first six months of the study, and then once every 6 months after that.
* Blood samples will be obtained in the first 5 days of treatment for pharmacokinetic studies and pharmacodynamic studies.
* Participants that are benefiting from the study treatment after the first cycle can continue to receive an additional 6 cycles of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* CLL/SLL with cells positive by flow cytometry (or immunostaining) for CD19, CD23, and CD5. Patients may be CD23 negative as long as they are also cyclin D1 negative or t(11;14) negative.
* Participants must have received at least 1 prior regimen containing a purine analogue or have received at least 2 chemotherapy regimens not containing a purine analogue. Patients may be refractory to single-agent purine analogue treatment, but patients may not be refractory to a combination of purine analogue with rituximab. Patients may have received rituximab.
* 18 years of age or older
* Able to take oral medications
* ECOG Performance Status of 2 or better
* Adequate organ function to tolerate chemotherapy
* Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the start of study drug administration and agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study is stopped.
* Require treatment based on 1996 NCI-WG criteria updated in 2008 by the IWCLL
* Patient agrees to discontinue St. John's Wort while receiving dasatinib therapy and stop at least 5 days before starting dasatinib.
* Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib

Exclusion Criteria:

* Pregnant or breastfeeding women
* Uncontrolled angina, congestive heart failure, or MI within 6 months
* Diagnosed or suspected congenital long QT syndrome
* Any history of clinically significant ventricular arrhythmias
* Prolonged QTc interval on pre-entry ECG
* Uncontrolled hypertension
* Hypokalemia or hypomagnesemia that is not corrected prior to dasatinib administration
* Patients should not be taking drugs that are generally accepted to have a risk of causing Torsades de Pointes
* Known HIV positive
* Known significant bleeding disorder unrelated to CLL
* Any significant pleural or pericardial effusion
* Patients may not have another malignancy that is uncontrolled or requires treatment within a year of starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Amrein, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
I do not plan to share IPD.

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib, Rituximab, Fludarabine: Single-arm
  dasatinib: Taken orally once a day on days 1-14 of each 28-day cycle
  Rituximab: Given intravenously, 375 mg/m2 each cycle (dose split, given on Days 3+4 of cycle 1, variable after that).
  fludarabine: Given intravenously, 25 mg/m2/day, for 3 doses per cycle (Days 3-5 in cycle 1, Days 1-3 after that)
Period: Overall Study
Arm/Group | Dasatinib, Rituximab, Fludarabine
Started | 10
Completed | 9
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib, Rituximab, Fludarabine
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 68 [60 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: To describe the response rate of complete response (CR) and partial response (PR) to treatment with this drug combination (SD=stable disease, PD=progressive disease)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib, Rituximab, Fludarabine
Number analyzed (Participants) | 10
Participants
  CR | 2
  PR | 2
  SD | 5
  PD | 1

2. Secondary Outcome: Progression-Free and Overall Survival
Description: To describe the progression-free and overall surivial
Time Frame: 2 years
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Dasatinib, Rituximab, Fludarabine
Number analyzed (Participants) | 10
months
  Progression-free survival | 8.75 [2.75 to 13]
  Overall survival | 24 [16.25 to 24]

3. Secondary Outcome: Toxicities
Description: Dasatinib may enhance the myelosuppression expected from fludarabine. This toxicity will be monitored with frequent CBC's. If after Day 21 of a cycle there is a grade 4 cytopenia, a dose reduction will occur in the next cycle of treatment, and that cycle cannot start until the ANC > 1,000 and the platelets > 25,000. There is also a risk for pleural effusions with dasatinib, but the risk will be low, since there is a break from dasatinib dosing on days 15-28 of each cycle. Nevertheless, if a grade 2 pleural effusion occurs, there will be a dose reduction in the next cycle of treatment.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib, Rituximab, Fludarabine
Number analyzed (Participants) | 10
Participants
  Platelets: 3 | 4
  Platelets: 4 | 3
  Platelets: 5 | 0
  Platelets: Did not have any | 3
  Neutropenia: 3 | 3
  Neutropenia: 4 | 3
  Neutropenia: 5 | 0
  Neutropenia: Did not have any | 4
  Fatigue: 3 | 1
  Fatigue: 4 | 0
  Fatigue: 5 | 0
  Fatigue: Did not have any | 9
  Dyspnea: 3 | 1
  Dyspnea: 4 | 0
  Dyspnea: 5 | 0
  Dyspnea: Did not have any | 9
  Pleural effusion: 3 | 1
  Pleural effusion: 4 | 0
  Pleural effusion: 5 | 0
  Pleural effusion: Did not have any | 9
  Bleeding: 3 | 1
  Bleeding: 4 | 0
  Bleeding: 5 | 0
  Bleeding: Did not have any | 9
  Fever alone: 3 | 1
  Fever alone: 4 | 0
  Fever alone: 5 | 0
  Fever alone: Did not have any | 9
  Infection: 3 | 0
  Infection: 4 | 0
  Infection: 5 | 1
  Infection: Did not have any | 9

ADVERSE EVENTS:
Arm/Group | Dasatinib, Rituximab, Fludarabine
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib, Rituximab, Fludarabine (N=10)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3, expected and possibly related
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 5, expected and possibly related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib, Rituximab, Fludarabine (N=10)
Fatigue (General disorders) | 5 (18)
Anemia (Blood and lymphatic system disorders) | 5 (14)
Platelet count decreased (Investigations) | 5 (14)
Nausea (Gastrointestinal disorders) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (12)
White blood cell decreased (Investigations) | 4 (11)
Blood bilirubin increased (Investigations) | 4 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Chills (General disorders) | 4 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (8)
Neutrophil count decreased (Investigations) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5)
Alkaline phosphatase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Edema limbs (General disorders) | 2 (3)
Mucosal infection (Infections and infestations) | 2 (3)
Lymphocyte count increased (Investigations) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (2)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Heart failure (Cardiac disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Gum infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Movements involuntary (Nervous system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Taste disturbance (Gastrointestinal disorders) | 1 (1)
Back- pain (General disorders) | 1 (1)
(General disorders) | 8 (10) — These events only had start and end dates entered but no information on the AE name or organ system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No